CLINICAL TRIAL: NCT02334592
Title: The Impact of Health Canada's Sunbed Exposure Time Guidelines on Serum 25(OH)D Concentrations
Brief Title: Vitamin D Production Levels Achieved by Sunbed Tanning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitamin D Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: VDS-1234
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: the effect of tanning; vitamin D production

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Pressure 100W sunbed (Experimental)
  Interventions: Radiation: Sunbed tanning
- Low Pressure 160W sunbed (Experimental)
  Interventions: Radiation: Sunbed tanning
- High Pressure sunbed (Experimental)
  Interventions: Radiation: Sunbed tanning
- Control group (No Intervention)

INTERVENTIONS:
Radiation: Sunbed tanning — Invention groups undergo a 12-week tanning protocol that follows Health Canada's RED Act
  Arms: High Pressure sunbed; Low Pressure 100W sunbed; Low Pressure 160W sunbed

SUMMARY:
Health Canada's Radiation Emitting Devices (RED) Act provides exposure time guidelines for sunbed use. These guidelines are intended to protect sunbed users from overexposure to UV radiation. Overexposure is defined as "exposure that exceeds the amount needed for vitamin D production and could lead to skin or eye damage. Acute overexposure induces sunburn." However, the effect of the recommended time exposure schedule on serum 25(OH)D response has not been characterized. Further, it is unknown if the maximum time exposures are required to reach and/or maintain optimal 25(OH)D levels. The aim of the current study is to characterize serum 25(OH)D response to regular sunbed use following the time exposure schedule recommended by Health Canada.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, male or female

Exclusion Criteria:

* History of skin cancer, granulomatous disease, liver disease, or kidney disease
* Photosensitive medications
* Pregnancy
* Vitamin D supplementation within last 60 days
* Sunbed use within last 60 days
* Planned travel to sunny destination during study period (January to April 2014)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To characterize serum 25(OH)D response to regular sunbed use, when performed according to the RED Act exposure time guidelines | 12 weeks

SECONDARY OUTCOMES:
To characterize serum 25(OH)D response with respect to sunbed lamp output (100W, 160W and High Pressure). | 12 weeks
To characterize serum 25(OH)D level with respect to skin lightness. | 12 weeks

REFERENCES:
- [Derived] Kimball SM, Lee J, Vieth R. Sunbeds with UVB radiation can produce physiological levels of serum 25-Hydroxyvitamin D in healthy volunteers. Dermatoendocrinol. 2017 Oct 17;9(1):e1375635. doi: 10.1080/19381980.2017.1375635. eCollection 2017. PMID 29484099